CLINICAL TRIAL: NCT00559052
Title: An Open-Label Cross-over Study to Evaluate the Intraduodenal Delivery of Lipase, Protease and Amylase From Administration of VIOKASE16 in Chronic Pancreatitis Subjects With Exocrine Pancreatic Insufficiency (EPI).
Brief Title: An Open-Label Study to Evaluate the Intraduodenal Delivery of Enzymes From Administration of VIOKASE16 in Exocrine Pancreatic Insufficiency (EPI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Axcan Pharma (Industry)
Collaborators: AAIPharma (Industry); Mayo Clinical Services (Unknown); City Hospital Laboratory Birmingham (Unknown)
Responsible Party: Jean Spenard/ Sr Dir, Clinical programs, Axcan Pharma
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: VIO16IP07-01
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Exocrine Pancreatic Insufficiency
Keywords: Enzymes; VIOKASE; Bioavailability
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Baseline measurement. No drug with the liquid meal during perfusion procedure to establish baseline secretion.
- 2 (Experimental): The Viokase 16 is to be taken as 3 tablets with the liquid meal during perfusion procedure.
  Interventions: Drug: VIOKASE 16

INTERVENTIONS:
Drug: VIOKASE 16 — The VIOKASE 16 is to be taken as 3 tablets with the perfusion procedure.
  Arms: 2

SUMMARY:
EPI leading to maldigestion is a frequent finding in many diseases of the pancreas, such as chronic pancreatitis (CP). Steatorrhea is the most important digestive manifestation in EPI. The current treatment of EPI includes enzyme supplementation with porcine pancreatic enzyme concentrate, consisting mainly of lipase, amylase and protease. An enzyme preparation able to deliver appropriate enzyme levels to the duodenum instead of the mid gut or distal small bowel, would appear to be clinically efficacious for the treatment of steatorrhea in subjects with CP suffering from EPI.

DETAILED DESCRIPTION:
Day of screening: Subjects will undergo screening procedures prior to entry into the study.

Day 0: Subjects will be admitted to the facility. Day 1: Subjects will undergo a first perfusion/aspiration procedure. Day 2: Subjects will rest. Day 3: Subjects will undergo a second perfusion/aspiration procedure. Day 4: Subjects will be discharged.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have the ability to give informed consent
* Female subjects must use a medically acceptable form of birth control and have a negative pregnancy test upon entering the study and not be breast-feeding
* Subjects must have medical condition compatible with exocrine pancreatic insufficiency
* Subjects must be off therapeutic doses of pancreatic enzyme supplementation prior to study entry day
* Subjects must be on omeprazole at least 5 days prior Day 0.

Exclusion Criteria:

* Subjects with a known hypersensitivity and/or contraindication to VIOKASE®16 or to any non-active component of VIOKASE or to any protein of porcine origin
* Subjects with a known hypersensitivity and/or contraindication to omeprazole or to any non-active component of omeprazole
* Subjects on enzyme therapy, H2-receptor antagonists, anticholinergics, antispasmodics prior to study entry
* Female subjects who are pregnant or lactating
* Subjects with acute pancreatitis or acute exacerbations of chronic pancreatic disease
* Subjects with a history of solid organ transplant or significant bowel resection between esophagus and pancreas
* Subjects who have received an investigational new drug within 30 days prior to entry into the study.
* Subjects with a known coagulopathy
* Subjects with any abnormal liver function test
* Subjects known to have a significant medical and/or mental disease that would compromise the subject's welfare or confound the study results
* Subjects who are not on omeprazole at least 5 days prior Day 0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Intraduodenal Lipase activity following single dose administration of VIOKASE16 tablets in EPI after a liquid meal. | 4 months

SECONDARY OUTCOMES:
Evaluation of the Intraduodenal protease and amylase activities following administration of VIOKASE16 tablets in EPI after a liquid meal. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Phillip P. Toskes, M.D., Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Shands Hospital, University of Florida, Gainesville, Florida
  - Santhi Swaroop Vege, M.D., Mayo Clinic- Rochester, Minnesota